CLINICAL TRIAL: NCT02599129
Title: An Exploratory Study to Evaluate the Safety and Efficacy of Secukinumab in the Treatment of Extensive Alopecia Areata
Brief Title: A Study of Secukinumab for the Treatment of Alopecia Areata
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Mark Lebwohl, Professor and System Chair, Dermatology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 15-0549
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata
MeSH Terms: conditions — Alopecia Areata | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Secukinumab (Experimental): 300 mg subcutaneous injections
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): matching placebo subcutaneous injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — subcutaneous secukinumab (300 mg) at weeks 0, 1, 2, 3, 4 and every 4 weeks thereafter up to and including Week 20.
  Arms: Secukinumab
Drug: Placebo — ￼subcutaneous placebo at weeks 0, 1, 2, 3, 4 and every 4 weeks thereafter up to and including week 20.
  Arms: Placebo

SUMMARY:
Alopecia areata is a medical condition, in which the hair falls out in patches. The hair can fall out on the scalp or elsewhere on the face and body.

Alopecia areata is an autoimmune skin disease, which means that the immune system is recognizing the hair follicles as foreign and attacking them, causing round patches of hair loss. It can progress to total scalp hair loss (alopecia totalis) or complete body hair loss (alopecia universalis). The scalp is the most commonly affected area, but the beard or any hair-bearing site can be affected alone or together with the scalp. Alopecia areata occurs in males and females of all ages, and is a highly unpredictable condition that tends to recur. Alopecia areata can cause significant distress to both patients and their families.

Aim: To assess the effects of a new treatment called secukinumab in patients with alopecia areata. A total of 30 patients will be included in the study, which will run for a total of 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years of age
* If female, the subject is not pregnant or nursing
* Subject is able to provide written informed consent and comply with the requirements of this study protocol.
* Subjects who are women of childbearing potential must have a negative urine pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 30 days before Day 0 and at least 6 months after the last study drug administration. Acceptable methods of birth control include intrauterine device (IUD); oral, transdermal, implanted or injected hormonal contraceptives (must have been initiated at least 1 month before entering the study); tubal ligation; abstinence and barrier methods with spermicide. Otherwise, if not of childbearing potential, subjects must: have a sterile or vasectomized partner; have had a hysterectomy, a bilateral oophorectomy or be clinically diagnosed infertile; or be in a menopausal state for at least a year.
* Subject with AA (unequivocal cases of AA), affecting at least 60% of the scalp, and present for at least 6 months.
* Tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) negative at the time of screening, or if patient has a history of positive PPD or QuantiFERON, he/she has completed the appropriate prophylaxis.
* Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, and physical examination.

Exclusion Criteria:

* Other concomitant types of alopecia (androgenetic, female pattern, traction, scarring and others)
* Any subject who is pregnant or refuses to practice an acceptable method of birth control (as stated in inclusion criterion # 4)
* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive tuberculin purified protein derivative (PPD) or QuantiFERON TB-Gold test (QFT) at screening. Subjects with a positive or indeterminate PPD or QFT test may participate in the study if a full tuberculosis work up (according to local practice/guidelines) is completed within 12 weeks prior to randomization and establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment must have been initiated at least for 4 weeks prior to randomization and the course of prophylaxis is planned to be completed.
* Active Crohn's disease
* Known hypersensitivity to latex
* Subjects with a history of HIV, or history of positive HCV or HBV
* Previous exposure to Secukinumab or other drug targeting IL-17A or its receptor; use of sensitizing therapy for alopecia areata including DPCP, squaric acid, DNCB within 1 month; PUVA, or any form of phototherapy within 1 month; use of any immunosuppressive therapies (systemic corticosteroids, methotrexate, azathioprine, mycophenolate mofetil, cyclosporine) within 1 month; or use of topical therapies (two weeks). All the above therapies will not be allowed during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from November 2015 to March 2016.
Groups:
- Placebo: Placebo: subcutaneous placebo at weeks 0, 1, 2, 3, 4 and every 4 weeks thereafter up to and including week 20.
Period: Overall Study
Arm/Group | Secukinumab | Placebo
Started | 7 | 4
Completed | 2 | 1
Not Completed | 5 | 3
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (14.3) | 52.2 (11.3) | 39.3 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Severity of Alopecial Tool (SALT) Score [Mean (Standard Deviation); unit: percent hair loss] — Scalp is divided into 4 areas namely, Vertex - 40% (0.4) of scalp surface area; right profile of scalp - 18% (0.18) of scalp surface area; left profile of scalp - 18% (0.18) of scalp surface area; Posterior aspect of scalp - 24% (0.24) of scalp surface area. Percentage of hair loss in any of these areas is percentage hair loss multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all above mentioned areas.
  percent hair loss
    SALT Score | 82.5 (19.3) | 95.3 (7.9) | 87.1 (8.6)
    Left profile of scalp | 83.6 (16.5) | 95.0 (10.0) | 87.7 (15.1)
    Right profile of scalp | 87.9 (12.9) | 95.0 (10.0) | 90.5 (11.9)
    Posterior profile of scalp | 84.3 (22.1) | 90.0 (14.1) | 86.4 (19.0)
    Vertex (Top) profile of scalp | 78.4 (27.2) | 98.75 (2.5) | 85.8 (23.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Severity of Alopecia Tool (SALT) Score of 50
Description: Number of subjects achieving a Severity of Alopecia Tool (SALT) score of 50 at Week 24
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

2. Secondary Outcome: Number of Subjects Achieving a SALT Score of 90 at Week 24
Description: We assessed the Number of subjects that achieved a SALT score of 90 at week 24
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

3. Secondary Outcome: Number of Subjects Achieving a SALT Score of 90 at Week 28
Description: We assessed the Number of subjects that achieved a SALT score of 90 at Week 28
Time Frame: week 28
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

4. Secondary Outcome: Number of Subjects Acheiving Physician's Global Assessment (PGA) Score of 3 or Above
Description: Number of subjects achieving a Physician's Global Assessment (PGA) score of 3 or above at week 24 (0, no regrowth; 1, <25% of regrowth; 2, 25%-49% of regrowth; 3, 50%-74% of regrowth; 4, 75%-99% of re- growth; 5, 100% of regrowth).
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

5. Secondary Outcome: Number of Subjects With Dermatology Life Quality Index (DLQI) of 3 or Above
Description: Number of subjects achieving a DLQI (Dermatology Life Quality Index), patient global assessment score of 3 or above at week 24 (0, no regrowth; 1, <25% of regrowth; 2, 25%-49% of regrowth; 3, 50%-74% of regrowth; 4, 75%-99% of re- growth; 5, 100% of regrowth).
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Secukinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 1/7 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Secukinumab (N=7) | Placebo (N=4)
Wisdom Tooth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Plaque Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes